CLINICAL TRIAL: NCT06337006
Title: Identification of Laryngeal Mask Airway Failure in Pediatric Patients With Objective Criteria: a Pilot Study
Brief Title: Laryngeal Mask Airway Failure in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SÜKAEK 2023/15/13
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Airway Management
Keywords: Laryngeal mask airway; pediatric; surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: The LMA was successfully placed after the first attempt.
  Interventions: Procedure: Placement of the laryngeal mask airway
- Group non-S: The LMA was not placed successfully after the first attempt.
  Interventions: Procedure: Placement of the laryngeal mask airway

INTERVENTIONS:
Procedure: Placement of the laryngeal mask airway — Evaluation of patients' chest movement with manual ventilation, airway leak level, airway pressures, fingertip O2 saturation percentage, and capnogram results will be recorded and the correlation between clinical observation and measured parameters will be evaluated.

SUMMARY:
There are a significant number of studies identifying risk factors for misplacement of LMAs. However, despite objective data indicating that tracheal intubation is performed inappropriately, such as air leaks, high air pressures, insufficient lung ventilation and single lung ventilation, which are easily identified after tracheal intubation, there are no objective data to define the misplacement of LMAs.

The aim of the study was to describe unsuccessful LMA placement in pediatric patients with objective data.

DETAILED DESCRIPTION:
Optimal use of extraglottic airways, including the laryngeal mask (LMA), has not been fully defined using real-world data. Usage patterns and the reported incidence of failure and complications in different geographic regions vary greatly. In the adult population, an observational study involving more than 15,000 cases revealed a 1.1% incidence of laryngeal mask failure, defined as intubation after laryngeal mask removal, and 62% of patients experienced significant airway complications.

Similar data are scarce in children. Pediatric laryngeal mask studies report adverse event frequencies ranging from 0% to 10%. These data are limited by the focus on specific surgical procedures or the small sample size resulting in simple univariate or inadequate multivariate analyses. Additionally, although data on adverse events are presented, laryngeal mask failure requiring endotracheal intubation has been reported infrequently.

There are a significant number of studies identifying risk factors for misplacement of LMAs. However, there are no objective data to define misplacement of LMAs.

1-2 mL of lidocaine gel was applied evenly to the classic LMA (Intavent Direct, Maidenhead, UK) capsule. The appropriate size of the LMA device (size 1.5 for 5-10 kg and size 2 for 10-20 kg) was selected according to the manufacturer's recommendation. The LMA was placed by an experienced anesthesiologist, with the patient's head in a neutral position, with a fully deflated cuff, and the patient's mouth was opened, then held parallel to the chest, and the device was advanced along the hard palate. The cuff of the device was inflated with a sufficient amount of air according to the manufacturer's instructions. After LMA placement, patients were divided into two groups as successful (Group S) or unsuccessful (Group non-S) according to bilateral equal chest movement during inspiration, square wave capnography, absence of gastric insufflation, epigastrium auscultation and adequate tidal volume delivery. Another experienced anesthesiologist recorded the set (8 mL/kg) tidal volume (VT), expiratory tidal volume, airway peak pressure, SpO2, EtCO2 measurements in three respiratory cycles. Airway leak (ΔVT); It was calculated by subtracting expiratory VT from the adjusted VT. Airway leak, airway peak pressure, SpO2 and EtCO2 measurement were determined as possible objective predictors for LMA placement failure. Postoperative airway complications; It was determined and recorded as soft tissue trauma, laryngospasm, bronchospasm, and severe cough attack.

The aim of the study was to describe unsuccessful LMA placement in pediatric patients with objective data.

ELIGIBILITY:
Inclusion Criteria:

* During surgery, the upper airway is planned to be supported with LMA by the Anesthesiologist.
* American Society of Anesthesiologists (ASA) physical status I or II

Exclusion Criteria:

* Surgery duration longer than 1 hour,
* Airway difficulty is expected,
* Restriction in opening the mouth,
* Airway malformation,
* Active upper respiratory tract infections,
* History of narrow airway,
* Hyperthyroidism, goiter, airway mass,
* Patients at risk of gastroesophageal reflux and aspiration of stomach contents

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children using a Laryngeal mask for airway control during surgery
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the unsuccess of placement of the laryngeal mask airway | 15 minute
  Identification of variables associated with unsuccessful LMA placement

SECONDARY OUTCOMES:
The relationship between LMA placement failure and postoperative airway complications | 2 hour
  Relationship between LMA placement failure with postoperative airway complications

CONTACTS AND LOCATIONS:
Overall Officials: OZGUR KOMURCU, 1, Study Director — Samsun University
Locations (1):
- Samsun University, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
non

REFERENCES:
- [Background] Farbood A, Tayyebi G, Naderi-Boldaji V, Asmarian N. Comparison of the ease of insertion and complications of the classical method of laryngeal mask airway insertion with an alternative method. Saudi J Anaesth. 2023 Apr-Jun;17(2):182-186. doi: 10.4103/sja.sja_681_22. Epub 2023 Mar 10. PMID 37260649
- [Background] Hernandez MR, Klock PA Jr, Ovassapian A. Evolution of the extraglottic airway: a review of its history, applications, and practical tips for success. Anesth Analg. 2012 Feb;114(2):349-68. doi: 10.1213/ANE.0b013e31823b6748. Epub 2011 Dec 16. PMID 22178627
- [Background] Van Zundert AAJ, Gatt SP, Kumar CM, Van Zundert TCRV, Pandit JJ. 'Failed supraglottic airway': an algorithm for suboptimally placed supraglottic airway devices based on videolaryngoscopy. Br J Anaesth. 2017 May 1;118(5):645-649. doi: 10.1093/bja/aex093. No abstract available. PMID 28510747